CLINICAL TRIAL: NCT00288613
Title: FREEDOM: Following Rehabilitation, Economics and Everyday-Dialysis Outcome Measurements Study
Status: Completed | Type: Observational
Sponsor: NxStage Medical (Other)
Responsible Party: Sponsor
Other Study IDs: CP0009
Record Dates: First submitted 2006-02-06; First posted 2006-02-08 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Kidney Failure, Chronic; End Stage Renal Disease, Requiring Dialysis
Keywords: ESRD; Daily Hemodialysis; Hemodialysis; Kidney Failure; Kidney Disease
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency; Kidney Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Purpose The purpose of this study is to compare the economical impact and clinical parameters of short daily hemodialysis using the NxStage® System One hemodialysis device with thrice-weekly conventional in-center dialysis using a matched cohort from the US Renal Data System (USRDS) database.

DETAILED DESCRIPTION:
In the 21st century, nephrologists in the United States face many challenges including a forecast of decline in physician manpower. Challenges that are specific to hemodialysis (HD) include reimbursement constraints, a growing shortage of nurses and major technological advances in dialysis equipment. There is a growing interest in alternative dialysis regimen and frequency, but a lack of patient incentive for self-care dialysis either in the center or in the home setting. The proposed phase 4 post-marketing study plans to explore whether daily HD is economically attractive compared with thrice weekly HD, while improving health-related quality of life and other dialysis adequacy measures. This project is unique as it provides a large prospective cohort of patients converted to daily HD, with a longitudinal follow up and an ability to compare to a matched cohort from the United States Renal Data Services. This study will help develop whether daily dialysis is economically attractive through the use of new technologies that reduce treatment costs and decrease hospitalization rates, with the long-term hope of increasing life expectancy. All patients will have the option to participate in the Quotidian Dialysis Registry, coordinated by the Lawson Health Research Institute (LHRI) in London, Ontario.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ESRD and require dialysis
* Medicare as primary payor (NOTE: Does not include Medicare HMO as primary payer)
* Candidate for daily hemodialysis (defined as 6 or more times per week)
* Ability to understand and willingness to sign an informed consent statement and a Health Insurance Portability and Accountability Act of 1996 (HIPAA) compliant authorization statement

Exclusion Criteria:

* Current use of the NxStage System One hemodialysis device
* Previous enrollment in this study
* Current enrollment in another investigational drug or device trial which might impact the outcome measures planned in this study
* Likelihood of not surviving the training period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with ESRD who are candidates for daily hemodialysis with the NxStage System One and have Medicare as the primary payor.
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2006-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Hospitalizations | duration of study participation
  To compare the all-cause hospitalizations reported in days per patient year on daily hemodialysis using NxStage System One hemodialysis device to thrice-weekly conventional in-center dialysis using a matched cohort from the US Renal Data System (USRDS) database

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand L. Jaber, MD, FASN, Principal Investigator — Unaffilated
Locations (41):
- United States (41):
  - Fort Smith Regional Dialysis Center, Fort Smith, Arkansas
  - Arkansas Nephrology Research Associates, Hot Springs, Arkansas
  - Renal Advantage (RAI), Garden Grove, California
  - Satellite Healthcare/Wellbound, Mountain View, California
  - Renal Advantage (RAI), Oakland, California
  - Kidney Center, Inc., Simi Valley, California
  - University of Colorado Hospital, Aurora, Colorado
  - Metabolism Associates - New Haven CAPD, New Haven, Connecticut
  - RAI Palm Harbor, Outcomes Research Int'l, Hudson, Florida
  - Emory, Renal Care Partners of Dunwoody, Sandy Springs, Georgia
  - Circle Medical Management, Chicago, Illinois
  - Affiliated Home Dialysis, Glen Ellyn, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Nephrology, Inc., Mishawaka, Indiana
  - Kansas Dialysis Services, Topeka, Kansas
  - University of Louisvile KDP, Louisville, Kentucky
  - Dialysis at Home, Inc, Brighton, Massachusetts
  - Great Lakes Renal Network, Alma, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Munson Dialysis Center, Traverse City, Michigan
  - Renal Advantage (RAI), Wyoming, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - NRA Home, Frontenac, Missouri
  - Washington University/Barnes Jewish Dialysis Center, St Louis, Missouri
  - Dialysis Center of Lincoln, Lincoln, Nebraska
  - Renal Advantage, Omaha, Nebraska
  - Silver Care Center, Cherry Hill, New Jersey
  - Lillian Booth Dialysis Center, Westwood, New Jersey
  - Apollo Healthcare - Niagara Renal Center, Niagara Falls, New York
  - Hortense and Louis Rubin Dialysis Center, Saratoga Springs, New York
  - Wake Forest University/Piedmont Dialysis, Winston-Salem, North Carolina
  - Community Physicians Dialysis Centers, Springfield, Ohio
  - Wellspan Dialysis, York, Pennsylvania
  - Renal Advantage (RAI), Charleston, South Carolina
  - Chattanooga Kidney Center, Chattanooga, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - Barlite SW Kidney Center, San Antonio, Texas
  - Renal Advantage (RAI), Hampton, Virginia
  - Virginia Commonwealth University/Medical College of Virginia, Richmond, Virginia
  - Northwest Kidney Centers, Seattle, Washington
  - Commonwealth Dialysis, Greenfield, Wisconsin

REFERENCES:
- [Derived] Cheetham MS, Ethier I, Krishnasamy R, Cho Y, Palmer SC, Johnson DW, Craig JC, Stroumza P, Frantzen L, Hegbrant J, Strippoli GF. Home versus in-centre haemodialysis for people with kidney failure. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD009535. doi: 10.1002/14651858.CD009535.pub3. PMID 38588450
- [Derived] Finkelstein FO, Schiller B, Daoui R, Gehr TW, Kraus MA, Lea J, Lee Y, Miller BW, Sinsakul M, Jaber BL. At-home short daily hemodialysis improves the long-term health-related quality of life. Kidney Int. 2012 Sep;82(5):561-9. doi: 10.1038/ki.2012.168. Epub 2012 May 23. PMID 22622497
- [Derived] Jaber BL, Schiller B, Burkart JM, Daoui R, Kraus MA, Lee Y, Miller BW, Teitelbaum I, Williams AW, Finkelstein FO; FREEDOM Study Group. Impact of short daily hemodialysis on restless legs symptoms and sleep disturbances. Clin J Am Soc Nephrol. 2011 May;6(5):1049-56. doi: 10.2215/CJN.10451110. Epub 2011 Mar 17. PMID 21415315
- [Derived] Jaber BL, Finkelstein FO, Glickman JD, Hull AR, Kraus MA, Leypoldt JK, Liu J, Gilbertson D, McCarthy J, Miller BW, Moran J, Collins AJ; FREEDOM Study Group. Scope and design of the Following Rehabilitation, Economics and Everyday-Dialysis Outcome Measurements (FREEDOM) Study. Am J Kidney Dis. 2009 Feb;53(2):310-20. doi: 10.1053/j.ajkd.2008.07.013. Epub 2008 Sep 27. PMID 18823688